CLINICAL TRIAL: NCT00978939
Title: Impact of Aggressive Versus Standard Drainage Regimen Using a Long Term Indwelling Pleural Catheter on the Incidence of Auto-Pleurodesis in Patients With Malignant Pleural Effusions
Brief Title: Impact of Aggressive Versus Standard Drainage Regimen Using a Long Term Indwelling Pleural Catheter
Acronym: ASAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00016092
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aggressive Drainage Arm (Experimental): Patients will drain up to 1 liter of pleural fluid everyday
  Interventions: Other: Aggressive Drainage Instructions
- Standard Drainage Arm (Active Comparator): Patients will drain up to 1 liter of pleural fluid every other day
  Interventions: Other: Standard Drainage Instructions

INTERVENTIONS:
Other: Standard Drainage Instructions — Patients will receive specific instructions to drain up to 1 liter of pleural fluid every other day
  Other Names: Conventional Drainage
  Arms: Standard Drainage Arm
Other: Aggressive Drainage Instructions — Patients will receive specific instructions to drain up to 1 liter of pleural fluid daily
  Other Names: Daily Drainage
  Arms: Aggressive Drainage Arm

SUMMARY:
Purpose and Objective: The purpose of this study is to determine if the rate of spontaneous pleurodesis using the Pleurx® catheter could be increased by simply increasing the frequency of pleural drainage and, if so, whether catheter-related complications can be minimized and spare patients the need for long term management of the Pleurx® catheter.

DETAILED DESCRIPTION:
Study Population: Patients greater than 18 years of age with malignant pleural effusions will be identified and approached in clinic by the Principle and Co-Investigator. Informed consent will be obtained from qualified and interested patients.

Study Activities: Patients will be randomized to standard and aggressive drainage groups and complete questionnaires regarding their health. Patients will then receive the Pleurx® catheter for standard treatment of their malignant pleural effusions, obtain a chest-xray, and receive educational instruction and training on catheter drainage and told whether to drain everyday using a 1-liter bottle or every other day using a 600-cc bottle. Patients will complete a drainage diary on everyday they drain fluid which will provide information on drainage volume, fluid color, pain, and complications. At 2 weeks, 6 weeks, and 12 weeks post catheter placement, patients will return to clinic for follow-up at which time they will have an interval history and physical and chest xray and complete a questionnaires regarding their health and satisfaction.

Risks/Safety Issues: Risks associated with draining the catheter include: pneumothorax, re-expansion pulmonary edema, hypotension, circulatory collapse, and infection. All serious adverse events will be reported to the institutional review board: a) death - immediately; b) life-threatening within 7 calendar days; c) all other SAEs (serious adverse events) within 15 calendar days. Should there be a serious adverse event that occurs that increases the risk to the participants, the study will be stopped, an investigation will be conducted, and a findings report will be generated before the study is resumed.

Data Analysis: The principal endpoint is the incidence of successful pleurodesis utilizing an aggressive drainage protocol compared to the incidence of successful pleurodesis using a standard drainage protocol. An interim analysis will be performed after 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years old
2. Pleural effusion (etiology fulfilling one of the following criteria):

   * Malignant effusion confirmed by cytology or pleural biopsy
   * Exudative effusion in the setting of known malignancy with no other identifiable cause
   * Malignant effusion due to tumors that are historically rapidly responsive to systemic therapy (small cell lung cancer, hematological malignancies) will only be included if refractory to standard chemotherapy
3. Symptoms such as shortness of breath, cough, or chest fullness/chest discomfort
4. Age greater than 18 years old
5. Pleural effusion (etiology fulfilling one of the following criteria):

   * Demonstration of symptomatic improvement after therapeutic thoracentesis (removal of ≤ 1.5 L of pleural fluid)
   * Recurrent pleural effusion after therapeutic thoracentesis

Exclusion Criteria:

1. Projected life expectancy less than 30 days as predicted by Karnofsky Performance Status score less than 30
2. Radiographic evidence of trapped lung - persistent lung collapse with failure of the lung to reexpand following drainage of a pleural effusion
3. Radiographic evidence of loculated pleural fluid
4. Previous attempted pleurodesis on the affected side
5. Previous lobectomy or pneumonectomy on the affected side
6. Patient receiving intrapleural chemotherapy
7. Chylothorax - pleural effusion with triglyceride levels > 110 mg/dl or chylomicrons on lipoprotein analysis, most commonly due to trauma/obstruction of the thoracic duct
8. Parapneumonic effusion - pleural effusion associated with pneumonia
9. Empyema - infected pleural space as defined by purulent pleural fluid, positive gram stain, or positive culture
10. Inability to adequately perform pleural drainage at home
11. Uncorrectable bleeding disorder
12. Skin infection at the site of intended catheter insertion
13. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-08; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of auto-pleurodesis utilizing aggressive drainage versus standard drainage protocols with the PleuRx® catheter | 2, 6, and 12 weeks post-catheter insertion

SECONDARY OUTCOMES:
To determine the median time to auto-pleurodesis utilizing aggressive drainage versus standard drainage protocols with the PleuRx® catheter | 2, 6, and 12 weeks post-catheter insertion
To assess the effects of aggressive drainage versus standard drainage protocols with the PleuRx® catheter on functional health status | 2, 6, and 12 weeks post-catheter insertion
To determine predictors of auto-pleurodesis (volume and rate of pleural fluid drainage, biochemical, and radiographic) using post-hoc analysis in both the aggressive and standard drainage protocols | 2, 6, and 12 weeks post-catheter insertion
To determine patient and caregivers' satisfaction with the PleuRx® catheter using a questionnaire | 2, 6, and 12 weeks post-catheter insertion

CONTACTS AND LOCATIONS:
Overall Officials: Momen Wahidi, MD, MBA, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - National Jewish Medical Center, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Tremblay A, Michaud G. Single-center experience with 250 tunnelled pleural catheter insertions for malignant pleural effusion. Chest. 2006 Feb;129(2):362-368. doi: 10.1378/chest.129.2.362. PMID 16478853
- [Background] Musani AI, Haas AR, Seijo L, Wilby M, Sterman DH. Outpatient management of malignant pleural effusions with small-bore, tunneled pleural catheters. Respiration. 2004 Nov-Dec;71(6):559-66. doi: 10.1159/000081755. PMID 15627865
- [Background] Barkauskas CE, Wahidi MM. Rate of auto pleurodesis with the indwelling pleural catheter using an aggressive drainage protocol in patients with malignant pleural effusions. Submitted for American Thoracic Society 2006 Meeting.